CLINICAL TRIAL: NCT02834416
Title: A Randomized Control Trial (RCT) and Economic Analysis of Two Exercise Delivery Methods in Men With Prostate Cancer on ADT
Brief Title: ADT Exercise Trial and Economic Analysis
Acronym: ADTExRCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Tom Baker Cancer Centre (Other); Southlake Regional Health Centre (Other); Scarborough Rouge Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-8158-CE
Record Dates: First submitted 2016-06-02; First posted 2016-07-15 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: An a priori decision was made to not include additional covariates in the ANCOVA model due to a smaller than anticipated sample size. Only trial centre, length of ADT, and baseline 6MWT will be included in the model.
  In addition, we have modified the wear time criteria for accelerometry from 600 minutes of wear time to 500 minutes of wear time. This allows for the inclusion of more participant data and more accurately reflects the clinical nature of this population.
  Amendment date: 17-Sep-20
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group-Supervised (Experimental): This intervention arm will include 3 group, supervised sessions per week for 6 months with a certified exercise specialist. Supervised sessions will be delivered in a group format with 4-8 participants per group. Flexibility training will include stretching for 5-10 minutes at the beginning and end of each session. Aerobic training will involve 30 minutes of low-impact step aerobics. Resistance training will be conducted using resistance bands, a stability ball, and an exercise mat with 8 prescribed exercises that target the major muscle groups. Participants will be encouraged to perform exercises independently on additional days, for a total of 4-5 days per week of exercise.
  Interventions: Behavioral: Supervised Group Exercise
- Home-Based (Experimental): The same protocol and training frequency as the supervised programs described above will be followed. However, all exercises will be completed independently by participants. Specific exercises in the aerobic program may be modified to accommodate patient preference (same target heart rate range as the supervised group). Participants will be supported with smartphone technology and remote 'health coaches' during the intervention phase. This will help to ensure participant adherence, appropriate progression, and safety.
  Interventions: Behavioral: Home Based Exercise

INTERVENTIONS:
Behavioral: Supervised Group Exercise — The exercise program will be delivered in a group format (4-8 participants per group) by a certified exercise specialist.
  Arms: Group-Supervised
Behavioral: Home Based Exercise — The exercise program will be executed independently by participants in a home-based setting. Home-based participants will be supported with remote health coaching and smartphone technology.
  Arms: Home-Based

SUMMARY:
Prostate Cancer (PC) affects 1 in 7 men. Nearly half of those diagnosed with PC will receive androgen deprivation therapy (ADT) as part of their treatment. ADT is good at managing PC but has many side effects. Researchers have shown that exercise, specifically one-on-one supervised exercise improves many of the side effects of ADT. However, exercise programs for men on ADT are not widely available. More questions need to be answered in order for exercise programs to become part of PC treatment. First, can programs that require fewer resources, such as group-exercise or home-based exercise, also improve ADT side-effects? Second, do exercise-related benefits continue beyond the structured exercise program? And what makes people continue exercising? Third, which exercise program is most cost-effective?

In this study, the investigators will compare: (a) group supervised in-centre and (b) home-based supported exercise programs to see which program is most effective for men with PC on ADT. The investigators will also look at what motivates people to continue to exercise both during a structured program and after the program is complete and will examine which exercise program is most cost-effective.

Participants (men with PC on ADT) will be recruited from one of the following cancer centres: Princess Margaret Cancer Centre in Toronto, the Tom Baker Cancer Centre in Calgary, the Southlake Regional Health Centre in Newmarket, and Scarborough and Rouge Hospital - Centenary Site in Scarborough. When a patient agrees to participate, patient will be randomly placed in 1 of 2 exercise programs. All programs will include the same type of exercises (aerobic, resistance and flexibility) and all participants will exercise 4-5 days per week for 30 minutes per day (as tolerated) for the length of the program (6 months). The investigators will look at how men with PC on ADT respond to the exercise program by measuring quality of life (QOL), fatigue and different physical measures before, during, and after the exercise program.

Although the investigators know that supervised one-on-one exercise is most effective at improving ADT side-effects, it is unknown if other forms of exercise are just as beneficial and more financially responsible. This study will allow the investigators to begin to answer these questions so that structured exercise programs become a regular part of PC treatment.

ELIGIBILITY:
Inclusion Criteria:

* men with histologically confirmed PC who are starting or continuing on ADT for at least 6 months or who are in an androgen-deprived (or castrate) state for the duration of the intervention
* fluent in English
* able to provide consent
* close to a study centre

Exclusion Criteria:

* already meeting guidelines for moderate to vigorous physical activity (MVPA) - conditions that would interfere with ability to participate

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-08; Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Fatigue (FACT-F) | Every 3 Months for 12 Months
  The FACT-F is a questionnaire that includes 13 items measuring cancer-related fatigue.
6 Minute Walk Test (6MWT) | Every 3 Months for 12 Months
  The 6MWT is a commonly used, validated measure that assesses functional endurance.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy-General (FACT-G) | Every 3 Months for 12 Months
  The FACT-G is a questionnaire that is well-validated and widely used to measure quality of life (QOL).
Functional Assessment of Cancer Therapy-Prostate (FACT-P) | Every 3 Months for 12 Months
  The FACT-P is a questionnaire that supplements the FACT-G with 12 prostate-specific items covering domains of urinary function, sexual function, pain, and related symptoms.
5 Times Sit to Stand Test | Every 3 Months for 12 Months
  A common, simple, and validated measure of functional lower body strength.
Grip Strength | Every 3 Months for 12 Months
  Grip strength is a measure of upper body strength and predicts long-term disability and mortality in middle-aged and older adults.
Bioelectrical Impedance Analysis | Every 6 Months for 12 Months
  Body composition will be measured using bioelectrical impedance analysis (BIA).
Waist Circumference and Hip Ratio | Every 6 Months for 12 Months
  Body composition will be measured using waist circumference(WC) and WC:hip ratio, following the standardized Canadian Society for Exercise Physiology - Physical Activity Training for Health (CSEP-PATH) protocol.
Body Mass Index | Every 6 Months for 12 Months
  Body composition will be measured using body mass index (BMI).
Bone Mineral Density (BMD) | Every 6 Months for 12 Months
  Bone mineral density will be measured at lumbar spine, hip, and distal 1/3 radius using dual x-ray absorptiometry (DXA).
Biological Outcomes (blood work) | Every 6 Months for 12 Months
  Fasting lipids, blood glucose, glycated hemoglobin, hemoglobin, prostate-specific antigen (PSA), and testosterone will be measured. Serum banking will also be done for use in future studies.
Sedentary Behaviour | Every 6 Months for 12 Months (unless otherwise specified)
  Time spent in activities that are characterized by an energy expenditure ≤ 1.5 metabolic equivalents and a sitting or reclining posture (sedentary behavior) will be assessed using the Sedentary Behaviour Questionnaire that is used in large cohort studies and has demonstrated evidence of reliability and validity.
Planning, Attitudes, & Barriers scale | Every 6 Months for 12 Months (unless otherwise specified)
  The Planning, Attitudes, & Barriers scale is a validated questionnaire that will be used to assess likelihood of exercise behavior over time.
Behavioral Regulations in Exercise Questionnaire-2 (BREQ-2) | Every 6 Months for 12 Months (unless otherwise specified)
  Behavioral Regulations in Exercise Questionnaire-2 (BREQ-2) is a validated questionnaire that assess predictors of adherence.
Psychological Need Support and Frustration Scale - Relatedness Items | Every 6 Months for 12 Months (unless otherwise specified)
  Relatedness will be assessed using the Psychological Need Support and Frustration Scale - Relatedness Items.
Health Care Climate Questionnaire (HCCQ) | Baseline only
  The Health Care Climate Questionnaire (HCCQ short form) assess participant perceptions of their health care team.
Walkability | Baseline only
  Participant postal codes will be collected to assess neighbourhood walkability (i.e., access to a grocery store within walking distance).
Disease-related Costs | Every 3 Months for 12 Months
  The investigators will collect economically relevant data about health status using preference-based (utility) instruments (European Quality of Life Five Dimensions Questionnaire, EQ-5D). Productivity losses and out-of-pocket expenditures, in addition to hospitalization, drug co-pay, and health visit data will be gathered using a patient questionnaire.
Exercise Adherence | Every 3 Months for 12 Months
  Both accelerometry and the Godin Leisure Time Exercise Questionnaire will be used as a measure of adherence at each time point. Both measures will provide a validated measure of physical activity.

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - University of Calgary/Tom Baker Cancer Centre, Calgary, Alberta
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Scarborough and Rouge Hospital, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alibhai SMH, Papadopoulos E, Mina DS, Ritvo P, Tomlinson G, Sabiston CM, Durbano S, Bremner KE, Chiarotto J, Matthew A, Warde P, O'Neill M, Culos-Reed SN. Home-based versus supervised group exercise in men with prostate cancer on androgen deprivation therapy: A randomized controlled trial and economic analysis. J Geriatr Oncol. 2024 Jan;15(1):101646. doi: 10.1016/j.jgo.2023.101646. Epub 2023 Nov 15. PMID 37976654
- [Derived] Alibhai SMH, Ritvo P, Santa Mina D, Sabiston C, Krahn M, Tomlinson G, Matthew A, Lukka H, Warde P, Durbano S, O'Neill M, Culos-Reed SN. Protocol for a phase III RCT and economic analysis of two exercise delivery methods in men with PC on ADT. BMC Cancer. 2018 Oct 23;18(1):1031. doi: 10.1186/s12885-018-4937-x. PMID 30352568